CLINICAL TRIAL: NCT01810172
Title: Digital Air Leak Monitoring for Patients Undergoing Lung Resection: A Randomized Controlled Clinical Trial
Brief Title: Digital Air Leak Monitoring for Patients Undergoing Lung Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Madelaine Plourde, Doctor, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-RS/2013-293
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Pneumothorax; Atelectasis
Keywords: lobectomy; segmentectomy; pneumothorax; pleural; digital; air leak
MeSH Terms: conditions — Pneumothorax; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry suction pleural drainage system (Active Comparator): The control group will have their chest tube connected to a dry suction pleural drainage system The intervention will be the dry suction pleural drainage system
  Interventions: Device: Dry suction pleura drainage device
- Digital pleural drainage system (Experimental): The experimental group will have their chest tube connected to a digital pleural drainage. The intervention will be the digital pleural drainage system.
  Interventions: Device: Digital pleural drainage system

INTERVENTIONS:
Device: Digital pleural drainage system — Reusable device with disposable collection system for digital monitoring of air leak.
  Other Names: ATMOS pleural drainage system
  Arms: Digital pleural drainage system
Device: Dry suction pleura drainage device — Disposable dry suction operating system. Collects pleural fluid and monitors for air leak.
  Other Names: Oasis dry suction water seal pleural drainage system
  Arms: Dry suction pleural drainage system

SUMMARY:
Often the decision for chest tube removal or trial of chest tube clamping is based on subjective assessment. This can lead to delay in chest tube removal. Recently, monitoring and recording of air leaks has been done using digital pleural drainage devices. This provides us with objective and continuous recording of air leaks as well as changes in pleural pressure. Our hypothesis is that the use of the ATMOS digital pleural drainage system will result in shorter hospital stay in comparison to traditional pleural drainage systems.

DETAILED DESCRIPTION:
Technology has become a driving force in surgery. From robotics to digital monitoring of oxygen saturation, it has revolutionized the way we care for patients. However, new technology comes at a cost to our healthcare system. It is therefore important to ensure that new devices actually improve outcomes. One example of this is minimally invasive surgery, which decreases morbidity to patients and reduces length of hospital stay. Unfortunately, despite this advance in lung surgery, delays in discharge from hospital are still prevalent due to prolonged air leaks. Many intra-operative methods have been explored in order to limit this issue with underwhelming success. This is why we are proposing a randomized controlled trial comparing a digital pleural collection system by ATMOS to traditional pleural collection devices by Atrium.

Our research question is: Can the use of a digital air leak monitoring system decrease hospital stay in patients undergoing anatomical lung resection when compared to traditional pleural drainage systems?

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 or older
* Patients undergoing a lobectomy or segmentectomy

Exclusion Criteria:

* Patients under the age of 18
* Patients undergoing pneumonectomy, wedge resection or bullectomy
* Patients who require additional procedures to control intraoperative air leak
* Patients who require mechanical ventilation post-operatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | one year
  The primary objective of this study will be the length of hospital stay from the day of surgery until the day of hospital discharge. The average length of hospital stay is 7 days.
  A subgroup analysis will be done to determine the impact of a video-assisted operative approach on length of stay and duration of chest tube drainage in comparison to thoracotomy.

SECONDARY OUTCOMES:
duration of chest tube insertion | one year
  The duration of chest tube drainage which will also be measured in days from the time of insertion in the operating room until they are removed.

OTHER OUTCOMES:
post chest tube removal complications | one year
  1. Post-chest tube removal pneumothorax. A significant pneumothorax will be defined as the presence of a space greater than 2cm at the apex and lateral aspect of the lung.
  2. Presence of atelectasis as determined by the dictating radiologist on chest x-ray from the second post-operative day.
  3. Need for chest tube re-insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Madelaine M Plourde, MD,MSc,FRCSC, Principal Investigator — CDHA
Locations (1):
- Capital Health District Authority, Halifax, Nova Scotia, Canada